CLINICAL TRIAL: NCT07252388
Title: Educational Intervention for Patient's Awareness on eaRly LDL-C Lowering Using Novel Pharmacological Strategies in secondarY Prevention (EARLY)
Brief Title: EARLY: Educational Intervention to Improve Patient Awareness on Early LDL-C Lowering in Secondary Prevention
Acronym: EARLY
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Heart Care Foundation (Other)
Collaborators: Novartis Farma S.p.A. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: K28
Record Dates: First submitted 2025-11-14; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Acute Coronary Syndromes; Chronic Coronary Syndromes
Keywords: educational intervention; Patient awareness; LDL cholesterol; Lipid lowering drugs; Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Intervention Model Description: Cluster randomized trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Quality-improvement educational intervention (Experimental): Patients included in the interventional arm will be guided to download a smartphone App which will allow them:
  * To see a 3-minute animated video aimed at explaining in layman terminology the benefits of intensifying LDL cholesterol reduction therapy, gaps in prescribing, reasons for clinical inertia, and motivations for patients to achieve recommended targets.
  * To see a check-list intended to propose a conscious way of managing dyslipidemia by the patient in relation to the targets to be achieved.
  * To include the ongoing lipid lowering therapy and enter the control LDL cholesterol value evaluated during hospitalization and that patient will perform in the days preceding the all the follow-up visits showing if goal has been achieved.
  Interventions: Other: Patient-oriented educational intervention
- Usual care (No Intervention): Patients followed in the centers randomized to the control arm will be managed by usual care in accordance with local clinical guidance.

INTERVENTIONS:
Other: Patient-oriented educational intervention — APP support
  Arms: Quality-improvement educational intervention

SUMMARY:
Cluster Randomized Trial to test the effectiveness of a patient level delivered educational intervention to improve the awareness on the relevance of obtaining LDL cholesterol recommended goals in patients admitted for an acute coronary syndrome, as compared to usual care. Overall, 24 sites (Coronary Care Units) will be included in the study, 12 randomized to the intervention and 12 to usual care. Overall, 240 patients will be enrolled during an acute coronary syndrome hospitalization.

DETAILED DESCRIPTION:
Elevated LDL cholesterol levels are associated with an increased risk of adverse events after an acute coronary syndrome. The higher the LDL cholesterol level at patients' admission for acute coronary syndrome, the greater the intensity of lipid-lowering treatment to be adopted to obtain the greatest benefits in terms of reduction of all-cause and cardiovascular mortality.

Despite European Society of Cardiology guideline recommendations to achieve low LDL cholesterol targets in patients with acute coronary syndrome (halving of baseline LDL cholesterol values and reaching LDL cholesterol values < 55 mg/dl or < 40 mg/dl in the case of a second event within two years of the first), this is unlikely to happen in clinical practice. Recent observational studies, such as the Da Vinci and Santorini, provide important insights into the practical management of lipid-lowering therapy in post-ACS patients in daily clinical practice, showing that only about 20% of high- or very-high-risk patients achieve guideline-recommended targets.

On the other hand, aggressive control of modifiable risk factors could prevent up to 80% of premature deaths related to cardiovascular disease. This underscores the importance of healthcare professionals in maximizing prevention efforts. Improvements in community health could prevent millions of serious cardiovascular events each year if properly implemented.

New therapies, such as PCSK9 inhibitors (monoclonal antibodies) or siRNA (inclisiran), offer an option for further and faster LDL cholesterol reduction during the peri- and post-acute coronary syndrome period, associated with a marked improvement in prognosis.

However, the use of these pharmacological strategies is currently quite limited in clinical practice. Several conditions account for the reduced "adherence" of clinicians and patients to the recommended therapies. Health disparities due to socioeconomic status, age, race, gender and cost, limited access to healthcare, perceived side effects associated with lipid-lowering therapies, health literacy and the presence of comorbidities, are all factors contributing to the suboptimal use of proposed therapies. Furthermore, clinical factors, including failure to identify patients requiring LDL cholesterol reassessment, insufficient monitoring, and clinical inertia have been associated with an insufficient use of lipid-lowering therapies.

Recently, the Italian Association of Hospital Cardiologists published a position paper on the treatment of hypercholesterolemia in patients with acute coronary syndrome. In the document, aimed at achieving the lipid targets outlined in the ESC/EAS 2019 guidelines more quickly than those currently recommended (from 8 weeks of the guidelines to 4 weeks of the Italian Association of Hospital Cardiologists document with a progressive and sustainable approach) and including new therapeutic options to reduce LDL cholesterol levels, a personalized therapeutic intervention based on LDL cholesterol levels at the time of hospital admission was proposed.

As a consequence, implementing lipid-lowering treatments early according to patients' clinical risk and the pharmacological options available to clinicians, while improving patients' awareness of cardiovascular risk, remains one of the primary objectives of the clinical cardiologist in secondary prevention.

Technology can effectively serve as an essential aid in achieving therapeutic targets. The introduction of dedicated applications could facilitate doctor-patient communication. On the basis of this evidence, the investigators designed the present study with the aim to evaluate if an educational intervention to improve the awareness on the relevance of obtaining LDL cholesterol recommended goals in patients with confirmed diagnosis of acute coronary syndrome, as compared to usual care can increase the proportion of patients at LDL cholesterol goal as suggested by 2019 ESC/EAS guidelines.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 and <80 years old.
2. Males and females at birth.
3. Baseline LDL-Cholesterol:

   * ≥ 130 mg/dl (in statin-naïve patients or who have not followed a stable (unchanged) statin regimen for at least 4 weeks prior to enrollment) or
   * ≥110 mg/dl (in patients who have received stable moderate-intensity or low-intensity statin treatment in the 4 weeks prior to enrollment) or
   * ≥100 mg/dl (in patients who have received stable treatment with high-intensity statins in the 4 weeks prior to enrollment)
4. Discharged at home
5. Ability to understand the requirements of the study and to provide informed consent

Exclusion Criteria:

1. Patients who have previously received or currently treated with PCSK9i (evolocumab or alirocumab) or siRNA (inclisiran)
2. Unstable clinical status (hemodynamic or electrical instability)
3. Uncontrolled cardiac arrhythmias, defined as recurrent, symptomatic ventricular tachycardia or atrial fibrillation or flutter with rapid ventricular response
4. Severe renal dysfunction, defined by eGFR < 30 mL/min/1.73 m2
5. Active liver disease or liver dysfunction, reported in the medical record or defined by AST or ALT levels > 3 times the upper limit of normal.
6. Reported intolerance to statins defined by the following criteria: inability to tolerate at least two different statins; intolerance associated with confirmed and intolerable statin-related adverse effects or significant biomarker abnormalities; improvement/resolution of symptoms or biomarkers following dose decrease or discontinuation; symptoms or changes in biomarkers not attributable to established predispositions.
7. Treatment with systemic steroids or systemic cyclosporine within the past 3 months (e.g., intravenously, intramuscularly, or orally)
8. Known active infection or severe hematologic, metabolic, or endocrine dysfunction as judged by the Investigator.
9. Current inclusion in other pharmacological and non-pharmacological experimental studies.
10. Pregnancy. For women of childbearing potential (age < 50 years and last menses <12 months prior to screening) who have not undergone tubal ligation, oophorectomy, or hysterectomy, pregnancy will be excluded from a pregnancy test prior to inclusion in the study.
11. Active neoplasia or very severe disease compromising short-medium term life expectancy.

Only for sites randomized to the interventional group:

• Patients without a device suitable for App use (eg. Smartphone or tablet) or patients that do not consent to receive push notifications by the App.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-12-11 (Estimated); Primary Completion 2027-08-11 (Estimated); Study Completion 2027-08-11 (Estimated)

PRIMARY OUTCOMES:
Number of patients achieving Guideline recommended LDL-Cholesterol goal | 12 month
  To compare the rate of patients with acute coronary syndrome who achieve the 2019 European Society of Cardiology/European Atherosclerosis Society guideline recommended LDL-Cholesterol goal (<55 mg/dl or <40 mg/dl in patients with recurrent events in the previous 24 months despite maximal lipid lowering treatment) at 12 months in sites following the interventional education protocol versus those receiving usual care.

SECONDARY OUTCOMES:
LDL-Cholesterol variation | 12 months
  Change in LDL-Cholesterol from baseline.
Use of Injective Lipid Lowering Therapy | 1 month
  Rate of patients who received PCSK9i inhibitors (monoclonal antibodies) or inclisiran during hospitalization (very fast track)
Use of Injective Lipid Lowering Therapy | 6 month
  Rate of patients who received PCSK9i inhibitors (monoclonal antibodies) or inclisiran during hospitalization (very fast track)
Number of participants with lipid lowering treatments related adverse events | 6 months
  In the eCRF at the 6-month follow-up visit discontinuation of lipid-lowering treatments will be recorded together with side effects most frequently associated with these treatments (e.g., arthralgia, limb pain, flu-like symptoms/malaise, myalgia, back pain, and elevated transaminases).
Number of participants with lipid lowering treatments related adverse events | 12 months
  In the eCRF at the 12-month follow-up visit discontinuation of lipid-lowering treatments will be recorded together with side effects most frequently associated with these treatments (e.g., arthralgia, limb pain, flu-like symptoms/malaise, myalgia, back pain, and elevated transaminases).

OTHER OUTCOMES:
Cardiovascular death (explorative objective) | 12 month
  Assess the rate of cardiovascular deaths
New hospitalizations for atherothrombotic events (explorative objective) | 12 month
  Assess the rate of new hospitalizations for atherothrombotic events.
All-cause mortality (explorative objective) | 12 month
  Assess the rate of all-cause mortality
All-cause hospitalizations (explorative objective) | 12 month
  Assess the rate of all-cause hospitalizations

CONTACTS AND LOCATIONS:
Locations (30):
- Italy (30):
  - AOU San Luigi Gonzaga - S.C.D.O. Cardiologia, Orbassano, TO
  - Ospedale Mauriziano Umberto I - SC Cardiologia, Torino, TO
  - Ospedale Miulli - U.O.C. Cardiologia - UTIC, Acquaviva delle Fonti
  - A.O.U. delle Marche - Cardiologia Ospedaliera e UTIC, Ancona
  - Ospedale Civile - U.O.C. di Cardiologia, Arzignano
  - Azienda Ospedaliera San Pio-PO G. Rummo - Cardiologia Interventistica e UTIC, Benevento
  - ARNAS G. Brotzu - Cardiologia con UTIC, Cagliari
  - Azienda Ospedaliera S. Anna e S. Sebastiano - U.O. Cardiologia d'Emergenza con UTIC, Caserta
  - Azienda Ospedaliera Cannizzaro - UOC Cardiologia, Catania
  - Ospedale Maggiore - U.O. Cardiologia e UTIC, Crema
  - PO S. Antonio Abate di Trapani - U.O.C. di Cardiologia, UTIC ed Emodinamica, Erice
  - Ospedale Padre Antero Micone - SC Cardiologia - UTIC, Genova
  - Ospedale Villa Scassi - ASL 3 Ligure - SC Cardiologia UTIC, Genova
  - Ospedali Riuniti - U.O.C. Cardiologia e UTIC, Livorno
  - ASST Ospedale Metropolitano Niguarda - Cardiologia 1 - Emodinamica, Milan
  - Fondazione IRCCS San Gerardo dei Tintori - Ospedale San Gerardo - U.O.C. Cardiologia, Monza
  - AORN Cardarelli - U.O. Cardiologia con UTIC, Napoli
  - AOR Villa Sofia-Cervello P.O. Cervello - U.O. Cardiologia - Cervello, Palermo
  - AOR Villa Sofia-Cervello PO Villa Sofia - UOC Cardiologia e UTIC e Emodinamica-Villa Sofia, Palermo
  - Fondazione IRCCS Policlinico San Matteo - UOC Cardiologia, Pavia
  - Ospedale Santo Spirito - Cardiologia con UTIC, Pescara
  - Ospedale Civile Guglielmo da Saliceto - UOC Cardiologia e UTIC, Piacenza
  - Ospedale Santo Stefano - U.O. Cardiologia, Prato
  - PO Santa Maria Nuova - AUSL RE IRCCS - SOC Cardiologia Ospedaliera, Reggio Emilia
  - P.O. San Filippo Neri - ASL ROMA 1 - Cardiologia Clinica e Riabilitativa, Roma
  - Ospedale San Camillo - UOC Cardiologia, Roma
  - Policlinico Casilino - U.O.C. Cardiologia, Roma
  - AOU S. Giovanni Di Dio-Ruggi D'Aragona - SSD UTIC, Salerno
  - Ospedale SS. Annunziata - Cardiologia Clinica ed Interventistica, Sassari
  - Ospedale Belcolle - UOSD UTIC Polo, Viterbo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] De Luca L, Riccio C, Navazio A, Valente S, Cipriani M, Corda M, De Nardo A, Francese GM, Napoletano C, Tizzani E, Roncon L, Caldarola P, Gulizia MM, Gabrielli D, Oliva F, Colivicchi F. ANMCO position paper on the management of hypercholesterolaemia in patients with acute coronary syndrome. Eur Heart J Suppl. 2023 May 18;25(Suppl D):D312-D322. doi: 10.1093/eurheartjsupp/suad100. eCollection 2023 May. PMID 37213800
- [Background] Mach F, Baigent C, Catapano AL, Koskinas KC, Casula M, Badimon L, Chapman MJ, De Backer GG, Delgado V, Ference BA, Graham IM, Halliday A, Landmesser U, Mihaylova B, Pedersen TR, Riccardi G, Richter DJ, Sabatine MS, Taskinen MR, Tokgozoglu L, Wiklund O; ESC Scientific Document Group. 2019 ESC/EAS Guidelines for the management of dyslipidaemias: lipid modification to reduce cardiovascular risk. Eur Heart J. 2020 Jan 1;41(1):111-188. doi: 10.1093/eurheartj/ehz455. No abstract available. PMID 31504418
- [Background] Ray KK, Molemans B, Schoonen WM, Giovas P, Bray S, Kiru G, Murphy J, Banach M, De Servi S, Gaita D, Gouni-Berthold I, Hovingh GK, Jozwiak JJ, Jukema JW, Kiss RG, Kownator S, Iversen HK, Maher V, Masana L, Parkhomenko A, Peeters A, Clifford P, Raslova K, Siostrzonek P, Romeo S, Tousoulis D, Vlachopoulos C, Vrablik M, Catapano AL, Poulter NR; DA VINCI study. EU-Wide Cross-Sectional Observational Study of Lipid-Modifying Therapy Use in Secondary and Primary Care: the DA VINCI study. Eur J Prev Cardiol. 2021 Sep 20;28(11):1279-1289. doi: 10.1093/eurjpc/zwaa047. PMID 33580789
- [Background] Ray KK, Haq I, Bilitou A, Manu MC, Burden A, Aguiar C, Arca M, Connolly DL, Eriksson M, Ferrieres J, Laufs U, Mostaza JM, Nanchen D, Rietzschel E, Strandberg T, Toplak H, Visseren FLJ, Catapano AL; SANTORINI Study Investigators. Treatment gaps in the implementation of LDL cholesterol control among high- and very high-risk patients in Europe between 2020 and 2021: the multinational observational SANTORINI study. Lancet Reg Health Eur. 2023 Apr 5;29:100624. doi: 10.1016/j.lanepe.2023.100624. eCollection 2023 Jun. PMID 37090089
- [Background] Byrne RA, Rossello X, Coughlan JJ, Barbato E, Berry C, Chieffo A, Claeys MJ, Dan GA, Dweck MR, Galbraith M, Gilard M, Hinterbuchner L, Jankowska EA, Juni P, Kimura T, Kunadian V, Leosdottir M, Lorusso R, Pedretti RFE, Rigopoulos AG, Rubini Gimenez M, Thiele H, Vranckx P, Wassmann S, Wenger NK, Ibanez B; ESC Scientific Document Group. 2023 ESC Guidelines for the management of acute coronary syndromes. Eur Heart J. 2023 Oct 12;44(38):3720-3826. doi: 10.1093/eurheartj/ehad191. No abstract available. PMID 37622654